CLINICAL TRIAL: NCT02578602
Title: MR Techniques in the Evaluation of Hepatocellular Carcinoma: Gadoxetate
Brief Title: MRI With Gadoxetate Disodium in Measuring Tumors in Patients With Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3L-10-1; NCI-2014-01850 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); USC 3L-10-1; HS-10-00188; 3L-10-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-09-13; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Adult Hepatocellular Carcinoma; Advanced Adult Hepatocellular Carcinoma; BCLC Stage 0 Adult Hepatocellular Carcinoma; BCLC Stage A Adult Hepatocellular Carcinoma; BCLC Stage B Adult Hepatocellular Carcinoma; BCLC Stage C Adult Hepatocellular Carcinoma; BCLC Stage D Adult Hepatocellular Carcinoma; Localized Non-Resectable Adult Liver Carcinoma; Localized Resectable Adult Liver Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — gadolinium ethoxybenzyl DTPA; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (gadoxetate disodium MRI) (Experimental): Patients receive gadoxetate disodium IV and then undergo enhanced liver MRI.
  Interventions: Drug: Gadoxetate Disodium; Device: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Gadoxetate Disodium — Given IV
  Other Names: Eovist; Gadolinium EOB DTPA; Gadolinium Ethoxybenzyl Diethylenetriaminepentaacetic Acid; Gadoxetic Acid Disodium; Gd-(S)-EOB-DTPA; Gd-EOB-DTPA; Primovist; ZK 139834
Device: Magnetic Resonance Imaging — Undergo MRI with gadoxetate disodium
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This pilot clinical trial studies magnetic resonance imaging (MRI) with gadoxetate disodium in measuring tumors in patients with liver cancer. Diagnostic procedures, such as MRI with gadoxetate disodium, may help find and diagnose liver cancer and find out how far the disease has spread. It is not yet known whether MRI with gadoxetate disodium provides a more precise measurement of liver tumors than standard computed tomography (CT).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the precision of gadoxetate (gadoxetate disodium)-enhanced MRI in evaluating lesion size.

II. To evaluate if there is a subjective improvement in the delineation of hepatocellular carcinoma (HCC) in the hepatocellular phase of contrast administration.

III. To further assess the sensitivity of gadoxetate-enhanced MRI for the detection of HCC.

SECONDARY OBJECTIVES:

I. To evaluate the reproducibility of various tumor measurement techniques in the evaluation of HCC.

II. To further evaluate how administration of gadoxetate affects diffusion weighted imaging.

OUTLINE:

Patients receive gadoxetate disodium intravenously (IV) and then undergo enhanced liver MRI.

After completion of study, patients are followed up at 2, 4, 8, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* CT features suggestive of HCC, including those features which have been described herein; they are also enumerated below:

  * For an arterially-enhancing lesion greater than or equal to 1 cm, but under 2 cm, all of the following criteria must be met:

    * Imaging features of a mass
    * Wash-out on later phases of contrast administration
    * At least 1 cm or more growth
  * For an arterially-enhancing lesion greater than or equal to 2 cm, two of the following criteria must be met:

    * Imaging features of a mass
    * Wash-out on later phases of contrast administration
    * At least 1 cm or more growth
  * All enhancing lesions with expansile, solid, enhancing tumor within vascular structures will be included, including the main portal vein, the main right and main left portal veins, the inferior vena cava (IVC), and the main hepatic veins
* No prior history of treatment of liver lesions
* Able to provide written and verbal informed consent
* Able to tolerate a complete abdominal MR examination, within 3 weeks of CT

Exclusion Criteria:

* Unable to provide written and verbal informed consent
* Unable to undergo MRI due to intraocular metallic foreign body, pacemaker, or other contraindications including objects in the body which are deemed to be unsafe or notable to be assessed, or unable to undergo MRI within 3 weeks of CT
* Pregnancy
* Severe renal insufficiency as defined by an estimated glomerular filtration rate of less than 30 cc/minute
* Severe liver disease as defined by Childs class C cirrhosis
* History of a previous reaction to contrast media
* History of bronchial asthma
* History of allergic disorders
* Acute renal insufficiency of any severity due to the hepato-renal syndrome or in the perioperative liver transplantation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-10; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Precision in tumor measurement for each type of image (CT vs. MRI), for each phase ( 4 for CT and 5 for MRI), and for each method of measuring "size" (1-,2-, and 3-dimensional), assessed by low inter- and intra-reader variability | Up to 24 hours
  Initially, a random effects analysis of variance (ANOVA) will be performed for each type of image (CT vs. MRI), for each phase (4 for CT and 5 for MRI) and for each method of measuring "size" (1-, 2-, and 3-dimensional) - for a total of 27 ANOVAs. Lesion, radiologist, and replication (for the 20 target lesions measured twice) will all be random effects; the inter-reader and the intra-reader variability will be estimated from these models and 95% confidence intervals will be constructed.

SECONDARY OUTCOMES:
Changes in apparent diffusion coefficient (ADC) values within lesions and within normal liver before and after administration of Gadoxetate | Up to 24 hours
  ADC values will be recorded for uninvolved liver parenchyma and for tumors before and after administration of gadoxetate disodium.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Whang, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States